CLINICAL TRIAL: NCT03567148
Title: Evaluation of The Effectiveness of Different Methods for Healing a Palatal Donor Site After Harvesting a Free Gingival Graft
Brief Title: The Effectiveness of Different Methods for Healing a Palatal Donor Site
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Sıla Çağrı İşler, Principal Investigator, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 36290600/114
Record Dates: First submitted 2018-05-16; First posted 2018-06-25 (Actual); Last update posted 2018-06-25 (Actual); Status verified 2018-06

CONDITIONS: Wound Heal; Graft Pain; Palate; Wound
Keywords: Graft; Pain; Palate; Wound healing
MeSH Terms: conditions — Wounds and Injuries; Pain | interventions — Equipment and Supplies; Low-Level Light Therapy; Collagen

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- PRF group (Active Comparator): Four layers of PRF membranes were placed in the palatal wound and sutured with 5/0 resorbable sutures
  Interventions: Procedure: PRF
- Essix retainer group (Active Comparator): An impression of palatal region was taken and the Essix retainer was prepared before the patients underwent surgery.
  Interventions: Procedure: Essix retainer
- Ozone therapy group (Active Comparator): Ozone was applied to the donor sites at five different points (four corner-points and a center point) at a fixed concentration of 2100 p.p.m. through a connected hand-piece, using a sterile, specially-formed perio-tip with 80% oxygen for 30 seconds. The applications were performed immediately after surgery and on the 1st, 3rd, and 7th days following the operation.
  Interventions: Procedure: Ozone therapy
- LLLT group (Active Comparator): Irradiation was performed at the same points described above using a diode laser (λ=970±15 nm, 14-W source power) (SIROLaser Xtend; Sirona Dental Systems GmbH, Bensheim, Germany) that continuously emitted a wavelength with 320µm fiberoptic; the power was 2W and the tissue dose was 35 J/cm2. Total irradiation time was 30 seconds. The applications were performed immediately after surgery, and on the 1st, 3rd and 7th, days following the operation.
  Interventions: Procedure: LLLT
- Collagen fleece group (Active Comparator): Collagen fleece (BEGO Collagen Fleece, Bremen, Germany) was sutured with 5/0 resorbable sutures (Pegesorb, Istanbul, Turkey) on the open wound with the aid of vertical mattress sutures.
  Interventions: Procedure: Collagen fleece
- Control group (No Intervention): Palatal wounds were left for spontaneous healing

INTERVENTIONS:
Procedure: PRF — Applying to the palatal wounds
  Other Names: medical device
  Arms: PRF group
Procedure: Essix retainer — Applying to the palatal wounds
  Other Names: medical device
  Arms: Essix retainer group
Procedure: Ozone therapy — Applying to the palatal wounds
  Other Names: medical device
  Arms: Ozone therapy group
Procedure: LLLT — Applying to the palatal wounds
  Other Names: medical device
  Arms: LLLT group
Procedure: Collagen fleece — Applying to the palatal wounds
  Other Names: medical device
  Arms: Collagen fleece group

SUMMARY:
Postoperative complications associated with free gingival graft (FGG) procedures are prolonged bleeding from the donor site, postoperative pain and delayed wound healing which increases the patients' morbidity. Hence, the aim of this study is to assess the effectiveness of different treatment modalities on palatal wound healing and patient's morbidity after FGG. Ninety patients requiring FGG were randomly will be assigned into six groups: group 1: Platelet rich fibrin (PRF) membrane, group 2: Essix retainer, group 3: topical ozone therapy, group 4: low-level laser therapy (LLLT), group 5: collagen fleece and group 6: untreated control group. Epithelization will be evaluated by means of bubble formation; sensitivity, edema, pain, changes in eating habits and burning sensation will be assessed by using visual analog scale (VAS) and also the presence of discomfort and bleeding will be evaluated in the postoperative first week and at 14 days, 1 and 3 months postoperatively.

DETAILED DESCRIPTION:
Inadequate attached gingiva is one of the major mucogingival problems for many individuals. However, the width of the keratinized tissue required to prevent periodontal disease remains unclear. Recently, a consensus report highlighted that if an individual's plaque control is suboptimal, a minimum of 2 mm of keratinized tissue and 1 mm of attached gingiva is needed.

Palatal keratinized mucosa is the most favorable donor region for a free gingival graft (FGG) due to its anatomic properties such as being histologically identical to keratinized attached mucosa of alveolar ridge and its ideal tissue thickness. The FGG surgical wound heals within 2-4 weeks, and prolonged bleeding, pain, and delayed wound healing of either the donor or recipient sites, which increases the patient's risk of morbidity, are the most common postoperative complications following surgery. Although homeostatic agents, mechanical barriers, and bioactive materials have been found to be effective in preventing these complications, the most ideal treatment has not yet been determined.

Platelet-rich fibrin (PRF), a platelet concentrate, is a safe and cost-effectiveness procedure that does not require biochemical blood handling. PRF has been used in many fields as an autologous biomaterial with a great healing potential for regenerating soft tissue and bones without inflammatory reactions, and it may be used to promote hemostasis and wound healing due to the presence of many growth factors. Recent studies have concluded that using PRF membranes after harvesting FGG enhances wound healing, reduces a patient's discomfort, and decreases need to change eating habits; thus, it reduces patient morbidity.

An Essix® retainer (Clear Advantage Series, Ortho Technology, Florida, USA) is a thermoplastic material used for stabilization after orthodontic treatment. It has been reported that gingival wounds that heal by secondary intention should be sheltered during the period of epithelization to protect against topical irritants, trauma, acidic or highly seasoned foods, and toothbrush abrasion.

It has been suggested that hemostatic agents provide faster and continuous hemostasis and make a positive contribution to early soft tissue healing. Application of hemostatic agents to the palatal donor sites has been found to be highly beneficial for achieving hemostasis in comparison to pressure only. Collagen fleece is a hemostatic agent that is made from the natural collagen of porcine dermis. The structure of the collagen promotes the formation and stabilization of blood clots during the initial wound healing phase. Recently, collagen-based materials have been used to improve early wound healing with an open healing design in the palatal area.

Ozone is a natural gaseous molecule made up of three oxygen atoms. The use of ozone has been proposed in dentistry because of its a strong oxidation effect and its antimicrobial potential, biocompatibility, and healing properties. In a previous study, the application of ozonated oil was reported to improve epithelial healing and gingival health following topical application. Taşdemir et al. concluded that ozone therapy could enhance wound healing, and the patients receiving this therapy experienced less pain after FGG operations than patients that had not received it.

Lower-level laser therapy (LLLT) is known as 'soft laser therapy' or 'bio-stimulation'. In dentistry, LLLT is usually used to accelerate wound healing, enhance remodeling and repair of bone, and reduce pain. Application of LLLT has been shown to improve wound healing after FGG and gingivectomy.

In light of this aforementioned information, it has been hypothesized that applications of PRF, an Essix retainer, collagen fleece, ozone therapy, and LLLT can result in improved wound healing after harvesting FGG in comparison to spontaneous healing. Thus, the present study aimed to assess and compare the effectiveness of these methods on palatal wound healing and patient morbidity.

ELIGIBILITY:
Inclusion Criteria:

* age >18,
* systemically healthy,
* non-smoker,
* full-mouth plaque and bleeding scores <20%,
* isolated gingival recession defects on the mandibular and maxillary anterior teeth with insufficient keratinized gingiva,

Exclusion Criteria:

* history of mucogingival surgery on the palatal area
* pregnancy
* systemic antibiotics taken for at least six months before the study
* having systemic diseases that could compromise wound healing

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
VAS questionnaire regarding to postoperative pain | 30th days postoperatively
  The VAS was divided into 10 segments, and the patients were asked to rank their pain level using a scoring system ranging from 0 to 10

SECONDARY OUTCOMES:
VAS questionnaire regarding to postoperative sensitivity | 30th days postoperatively
  The VAS was divided into 10 segments, and the patients were asked to rank their sensitivity level using a scoring system ranging from 0 to 10
hydrogen peroxide test | 30th days postoperatively
  Epithelization was evaluated using the same time-points by means of bubble formation after dripping hydrogen peroxide (3%) onto the operation site
VAS questionnaire regarding to changes in eating habits | 30th days postoperatively
  The VAS was divided into 10 segments, and the patients were asked to rank their eating habits level using a scoring system ranging from 0 to 10
VAS questionnaire regarding to burning sensation | 30th days postoperatively
  The VAS was divided into 10 segments, and the patients were asked to rank their sense of burning level using a scoring system ranging from 0 to 10

CONTACTS AND LOCATIONS:
Overall Officials: Deniz Cetiner, Prof. Dr., Study Director — Gazi University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gumus P, Buduneli E. Graft stabilization with cyanoacrylate decreases shrinkage of free gingival grafts. Aust Dent J. 2014 Mar;59(1):57-64. doi: 10.1111/adj.12149. Epub 2014 Feb 4. PMID 24494804
- [Background] Harrison JS, Conlan MJ, Deas DE. An alternative donor site for an epithelialized-free soft-tissue autograft. Compend Contin Educ Dent. 2011 Mar;32(2):e29-31. PMID 23738833
- [Background] Kim DM, Neiva R. Periodontal soft tissue non-root coverage procedures: a systematic review from the AAP Regeneration Workshop. J Periodontol. 2015 Feb;86(2 Suppl):S56-72. doi: 10.1902/jop.2015.130684. PMID 25644300
- [Background] Sanz M, Simion M; Working Group 3 of the European Workshop on Periodontology. Surgical techniques on periodontal plastic surgery and soft tissue regeneration: consensus report of Group 3 of the 10th European Workshop on Periodontology. J Clin Periodontol. 2014 Apr;41 Suppl 15:S92-7. doi: 10.1111/jcpe.12215. PMID 24641004
- [Background] Brasher WJ, Rees TD, Boyce WA. Complications of free grafts of masticatory mucosa. J Periodontol. 1975 Mar;46(3):133-8. doi: 10.1902/jop.1975.46.3.133. PMID 1079047
- [Background] Keceli HG, Aylikci BU, Koseoglu S, Dolgun A. Evaluation of palatal donor site haemostasis and wound healing after free gingival graft surgery. J Clin Periodontol. 2015 Jun;42(6):582-9. doi: 10.1111/jcpe.12404. Epub 2015 May 19. PMID 25892528
- [Background] Dohan DM, Choukroun J, Diss A, Dohan SL, Dohan AJ, Mouhyi J, Gogly B. Platelet-rich fibrin (PRF): a second-generation platelet concentrate. Part I: technological concepts and evolution. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2006 Mar;101(3):e37-44. doi: 10.1016/j.tripleo.2005.07.008. Epub 2006 Jan 19. PMID 16504849
- [Background] Borie E, Olivi DG, Orsi IA, Garlet K, Weber B, Beltran V, Fuentes R. Platelet-rich fibrin application in dentistry: a literature review. Int J Clin Exp Med. 2015 May 15;8(5):7922-9. eCollection 2015. PMID 26221349
- [Background] Kulkarni MR, Thomas BS, Varghese JM, Bhat GS. Platelet-rich fibrin as an adjunct to palatal wound healing after harvesting a free gingival graft: A case series. J Indian Soc Periodontol. 2014 May;18(3):399-402. doi: 10.4103/0972-124X.134591. PMID 25024559
- [Background] Femminella B, Iaconi MC, Di Tullio M, Romano L, Sinjari B, D'Arcangelo C, De Ninis P, Paolantonio M. Clinical Comparison of Platelet-Rich Fibrin and a Gelatin Sponge in the Management of Palatal Wounds After Epithelialized Free Gingival Graft Harvest: A Randomized Clinical Trial. J Periodontol. 2016 Feb;87(2):103-13. doi: 10.1902/jop.2015.150198. Epub 2015 Aug 27. PMID 26313017
- [Background] Rossmann JA, Rees TD. A comparative evaluation of hemostatic agents in the management of soft tissue graft donor site bleeding. J Periodontol. 1999 Nov;70(11):1369-75. doi: 10.1902/jop.1999.70.11.1369. PMID 10588501
- [Background] Silverstein ME, Chvapil M. Experimental and clinical experiences with collagen fleece as a hemostatic agent. J Trauma. 1981 May;21(5):388-93. doi: 10.1097/00005373-198105000-00011. PMID 7230285
- [Background] Thoma DS, Hilbe M, Bienz SP, Sancho-Puchades M, Hammerle CH, Jung RE. Palatal wound healing using a xenogeneic collagen matrix - histological outcomes of a randomized controlled clinical trial. J Clin Periodontol. 2016 Dec;43(12):1124-1131. doi: 10.1111/jcpe.12624. Epub 2016 Oct 25. PMID 27616435
- [Background] Nogales CG, Ferrari PH, Kantorovich EO, Lage-Marques JL. Ozone therapy in medicine and dentistry. J Contemp Dent Pract. 2008 May 1;9(4):75-84. PMID 18473030
- [Background] Patel PV, Kumar V, Kumar S, Gd V, Patel A. Therapeutic effect of topical ozonated oil on the epithelial healing of palatal wound sites: a planimetrical and cytological study. J Investig Clin Dent. 2011 Nov;2(4):248-58. doi: 10.1111/j.2041-1626.2011.00072.x. Epub 2011 Jul 7. PMID 25426896
- [Background] Tasdemir Z, Alkan BA, Albayrak H. Effects of Ozone Therapy on the Early Healing Period of Deepithelialized Gingival Grafts: A Randomized Placebo-Controlled Clinical Trial. J Periodontol. 2016 Jun;87(6):663-71. doi: 10.1902/jop.2016.150217. Epub 2016 Jan 16. PMID 26777769
- [Background] Aggarwal H, Singh MP, Nahar P, Mathur H, Gv S. Efficacy of low-level laser therapy in treatment of recurrent aphthous ulcers - a sham controlled, split mouth follow up study. J Clin Diagn Res. 2014 Feb;8(2):218-21. doi: 10.7860/JCDR/2014/7639.4064. Epub 2014 Feb 3. PMID 24701539
- [Background] Ustaoglu G, Ercan E, Tunali M. Low-Level Laser Therapy in Enhancing Wound Healing and Preserving Tissue Thickness at Free Gingival Graft Donor Sites: A Randomized, Controlled Clinical Study. Photomed Laser Surg. 2017 Apr;35(4):223-230. doi: 10.1089/pho.2016.4163. Epub 2017 Jan 12. PMID 28092488
- [Background] Ozcelik O, Cenk Haytac M, Kunin A, Seydaoglu G. Improved wound healing by low-level laser irradiation after gingivectomy operations: a controlled clinical pilot study. J Clin Periodontol. 2008 Mar;35(3):250-4. doi: 10.1111/j.1600-051X.2007.01194.x. PMID 18269665